CLINICAL TRIAL: NCT02015793
Title: A Phase 2, Randomized, Double-Blind, Multicenter Study to Evaluate the Pharmacokinetics, Safety, and Efficacy of Two Adalimumab Dosing Regimens in Chinese Subjects With Moderately to Severely Active Crohn's Disease and Elevated High-Sensitivity C-reactive Protein
Brief Title: Study to Evaluate the Pharmacokinetics, Safety and Efficacy of Two Treatment Modules in Chinese Subjects With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M14-232
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2016-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Pharmacokinetics
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Induction Dose (Experimental): Participants received the low loading dose of adalimumab (80 mg at Week 0) followed by the standard maintenance dose of adalimumab (40 mg every other week) at Weeks 2, 4, and 6.
  Interventions: Biological: Adalimumab; Biological: Placebo for adalimumab
- Standard Induction Dose (Experimental): Participants received the standard loading dose of adalimumab (160 mg at Week 0 and 80 mg at Week 2) followed by the standard maintenance dose of adalimumab (40 mg every other week) at Weeks 4 and 6.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous injection.
Biological: Placebo for adalimumab — Placebo for adalimumab pre-filled syringe, administered by subcutaneous injection to maintain double-blind.
  Arms: Low Induction Dose

SUMMARY:
The purpose of this study is to investigate the efficacy, safety, and pharmacokinetics of adalimumab following subcutaneous (SC) administration of 2 dosing regimens in Chinese subjects with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of Chinese descent with full Chinese parentage.
2. Diagnosis of Crohn's disease (CD) for at least 3 months prior to Week 0 confirmed by endoscopy, radiologic evaluation, and/or histology during the Screening Period.
3. Crohn's Disease Activity Index (CDAI) ≥ 220 and ≤ 450 despite treatment with oral corticosteroids and/or immunosuppressants.
4. Subject has a negative Tuberculosis (TB) Screening Assessment.

Exclusion Criteria:

1. Subject with ulcerative colitis or indeterminate colitis.
2. Subject who has had a surgical bowel resection within the past 6 months or who is planning any resection at any time point in the future.
3. Subject with an ostomy or ileoanal pouch.
4. Subject who has short bowel syndrome.
5. Subject with symptomatic known obstructive strictures.
6. Subject with an internal or external fistula (with the exception of an anal fistula without abscess).
7. Chronic recurring infections or active TB.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Robinson, Study Director — AbbVie

REFERENCES:
- [Result] Wu KC, Ran ZH, Gao X, Chen M, Zhong J, Sheng JQ, Kamm MA, Travis S, Wallace K, Mostafa NM, Shapiro M, Li Y, Thakkar RB, Robinson AM. Adalimumab induction and maintenance therapy achieve clinical remission and response in Chinese patients with Crohn's disease. Intest Res. 2016 Apr;14(2):152-63. doi: 10.5217/ir.2016.14.2.152. Epub 2016 Apr 27. PMID 27175116
- See also: Related Info. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Induction Dose | Standard Induction Dose
Started | 15 | 15
Completed Double-Blind Period | 14 | 14
Entered Open-label Extension Period | 13 | 14
Completed | 11 | 11
Not Completed | 4 | 4
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Induction Dose | Standard Induction Dose | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (14.60) | 35.6 (13.00) | 34.5 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Serum Adalimumab Concentration at Week 8
Description: Blood samples were drawn prior to drug administration. Adalimumab concentrations in serum were determined using a validated enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Week 8
Population: All participants in the intent-to-treat (ITT) population, defined as all randomized participants who received at least 1 dose of double-blind study drug, who had evaluable data.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 14 | 12
μg/mL | 7.99 (3.48) | 10.0 (4.57)

2. Secondary Outcome: Number of Participants With Potentially Significant Hematology Parameters During Administration of Adalimumab
Description: The number of participants with an abnormal laboratory result meeting Common Toxicity Criteria (CTC) Version 3.0 (or later) of Grade 3 or higher is summarized. n=the number of participants with CTC Grade <3 at baseline and a post-baseline value for each parameter.
Time Frame: 26 weeks
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 15 | 15
participants
  Haemoglobin <80 g/L (n=15,15) | 1 | 1
  White Blood Cells ≥1 x10^9/L (n=15,15) | 1 | 0
  Neutrophils <1.0x10^9/mcL (n=15,15) | 1 | 0
  Lymphocytes <0.5x10^3/mcL (n=15,13) | 2 | 0

3. Secondary Outcome: Number of Participants With Potentially Significant Clinical Chemistry Parameters During Administration of Adalimumab
Description: The number of participants with an abnormal laboratory result meeting Common Toxicity Criteria (CTC) Version 3.0 (or later) of Grade 3 or higher is summarized.
Time Frame: From Week 0 to Week 26
Population: Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 15 | 15
participants
  Potassium <3.0 mmol/L | 0 | 1
  Sodium <130 mmol/L | 0 | 1
  Albumin <20 g/L | 0 | 1
  Calcium <1.75 mmol/L | 0 | 1
  Uric Acid >500µmol/L | 0 | 1

4. Secondary Outcome: Number of Participants With Potentially Significant Vital Signs Parameters During Administration of Adalimumab
Description: Blood pressure and pulse were measured while the participant was sitting. The number of participants with a postbaseline vital sign result that meets Common Toxicity Criteria (CTC) version 3.0 (or later) Grade 3 or higher and is also more extreme than the baseline value is summarized. Terms abbreviated in the table include systolic blood pressure (SBP) and diastolic blood pressure (DBP). Increase and decrease are signified by ↑ and ↓, respectively.
Time Frame: 26 weeks
Population: Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 15 | 15
participants
  SBP ≤90 mm Hg or ≥20 mm Hg ↓ from BL | 7 | 5
  SBP ≥180 mm Hg or ≥20 mm Hg ↑ from BL | 8 | 3
  DBP ≤50 mm Hg or ≥15 mm Hg ↓ from BL | 3 | 4
  SBP ≥105 mm Hg or ≥15 mm Hg ↑ from BL | 6 | 4
  Pulse ≤50 bpm or ≥15 bpm ↓ from BL | 6 | 7
  Pulse SBP ≥120 bpm or ≥15 bpm ↑ from BL | 7 | 6

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant which does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs or TESAE) are defined as any event that began or worsened in severity after the first dose of study drug. The investigator assessed the relationship of each event to the use of study drug as either Reasonable possibility or No reasonable possibility of being related to study drug.
  For more details on adverse events please see the AE section below.
Time Frame: 35 weeks
Population: Safety Analysis Set.
Measure: Number; unit: participants
Groups:
- Low Induction Dose (Double-blind Period): Participants received the low loading dose of adalimumab (80 mg at Week 0) followed by the standard maintenance dose of adalimumab (40 mg every other week) at Weeks 2, 4, and 6.
- Standard Induction Dose (Double-blind Period): Participants received the standard loading dose of adalimumab (160 mg at Week 0 and 80 mg at Week 2) followed by the standard maintenance dose of adalimumab (40 mg every other week) at Weeks 4 and 6.
- Low Induction Dose (Open-label Extension Period); Standard Induction Dose (Open-label Extension): Participants received open-label adalimumab 40 mg every other week for 18 weeks.
Arm/Group | Low Induction Dose (Double-blind Period) | Standard Induction Dose (Double-blind Period) | Low Induction Dose (Open-label Extension Period) | Standard Induction Dose (Open-label Extension)
Number analyzed (Participants) | 15 | 15 | 13 | 14
participants
  Any TEAE | 6 | 7 | 7 | 7
  Any TESAE | 1 | 1 | 1 | 2
  TEAE leading to discontinuation | 2 | 1 | 1 | 2
  Severe TEAE | 0 | 1 | 0 | 1
  TEAEs with reasonable possibility of being related | 3 | 6 | 5 | 6
  Deaths | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission (Crohn's Disease Activity Index [CDAI] < 150) Every 2 Weeks up to Week 26
Description: CDAI is used to quantify the signs and symptoms of patients with Crohn's Disease. A score below 150 indicates remission and a score of 220 to 450 reflects moderate to severe disease. Non-responder imputation (NRI) for missing CDAI observations was used.
Time Frame: Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 15 | 15
percentage of participants
  Week 2 | 26.7 [7.8 to 55.1] | 46.7 [21.3 to 73.4]
  Week 4 | 40.0 [16.3 to 67.7] | 66.7 [38.4 to 88.2]
  Week 6 | 60.0 [32.3 to 83.7] | 73.3 [44.9 to 92.2]
  Week 8 | 60.0 [32.3 to 83.7] | 66.7 [38.4 to 88.2]
  Week 10 | 66.7 [38.4 to 88.2] | 66.7 [38.4 to 88.2]
  Week 12 | 60.0 [32.3 to 83.7] | 73.3 [44.9 to 92.2]
  Week 14 | 60.0 [32.3 to 83.7] | 73.3 [44.9 to 92.2]
  Week 16 | 60.0 [32.3 to 83.7] | 73.3 [44.9 to 92.2]
  Week 18 | 60.0 [32.3 to 83.7] | 73.3 [44.9 to 92.2]
  Week 20 | 66.7 [38.4 to 88.2] | 66.7 [38.4 to 88.2]
  Week 22 | 66.7 [38.4 to 88.2] | 66.7 [38.4 to 88.2]
  Week 24 | 66.7 [38.4 to 88.2] | 66.7 [38.4 to 88.2]
  Week 26 | 66.7 [38.4 to 88.2] | 66.7 [38.4 to 88.2]

7. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response (CDAI Decrease ≥ 70 From Week 0) Every 2 Weeks up to Week 26
Description: as for outcome 6
Time Frame: Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 15 | 15
percentage of participants
  Week 2 | 66.7 [38.4 to 88.2] | 80.0 [51.9 to 95.7]
  Week 4 | 93.3 [68.1 to 99.8] | 93.3 [68.1 to 99.8]
  Week 6 | 93.3 [68.1 to 99.8] | 86.7 [59.5 to 98.3]
  Week 8 | 93.3 [68.1 to 99.8] | 86.7 [59.5 to 98.3]
  Week 10 | 86.7 [59.5 to 98.3] | 86.7 [59.5 to 98.3]
  Week 12 | 80.0 [51.9 to 95.7] | 80.0 [51.9 to 95.7]
  Week 14 | 73.7 [44.9 to 92.2] | 73.7 [44.9 to 92.2]
  Week 16 | 80.0 [51.9 to 95.7] | 73.7 [44.9 to 92.2]
  Week 18 | 80.0 [51.9 to 95.7] | 73.7 [44.9 to 92.2]
  Week 20 | 73.7 [44.9 to 92.2] | 66.7 [38.4 to 88.2]
  Week 22 | 66.7 [38.4 to 88.2] | 66.7 [38.4 to 88.2]
  Week 24 | 66.7 [38.4 to 88.2] | 66.7 [38.4 to 88.2]
  Week 26 | 66.7 [38.4 to 88.2] | 66.7 [38.4 to 88.2]

8. Secondary Outcome: CDAI: Mean Change From Baseline to Each Visit
Description: CDAI is used to quantify the signs and symptoms of patients with Crohn's Disease. Scores range from 0 to approximately 600. A score below 150 indicates remission and a score of 220 to 450 reflects moderate to severe disease. Last observation carried forward (LOCF) for missing CDAI observations was used.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 15 | 15
units on a scale
  Week 2 | -108.91 (76.196) | -143.79 (86.193)
  Week 4 | -152.96 (71.589) | -163.21 (95.545)
  Week 6 | -163.53 (80.868) | -178.23 (103.159)
  Week 8 | -181.50 (81.611) | -181.87 (100.077)
  Week 10 | -185.24 (81.532) | -182.87 (96.039)
  Week 12 | -200.33 (88.612) | -191.09 (98.035)
  Week 14 | -193.63 (97.130) | -194.96 (111.444)
  Week 16 | -198.07 (96.381) | -191.37 (108.932)
  Week 18 | -200.17 (93.758) | -188.31 (109.516)
  Week 20 | -214.43 (96.417) | -189.83 (110.845)
  Week 22 | -213.95 (98.357) | -194.53 (111.046)
  Week 24 | -215.47 (99.278) | -187.98 (107.702)
  Week 26 | -215.79 (101.879) | -200.17 (110.999)

9. Secondary Outcome: High-sensitivity C-reactive Protein (hsCRP): Median Change From Baseline (Week 0) to Week 26
Description: hsCRP was measured from blood samples as a marker for inflammation. Higher levels are indicative of more inflammation. Normal concentration in healthy human serum is usually lower than 3 mg/L, slightly increasing with age. LOCF was used for missing data.
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, and 26
Population: ITT population.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 15 | 15
mg/L
  Week 1 | -7.70 [-74.8 to 28.1] | -24.51 [-187.6 to -1.7]
  Week 2 | -14.10 [-83.3 to 32.3] | -25.37 [-184.7 to 5.3]
  Week 4 | -12.05 [-93.2 to 42.2] | -21.12 [-170.6 to 43.0]
  Week 6 | -12.66 [-94.6 to 46.2] | -21.61 [-165.9 to 18.2]
  Week 8 | -11.90 [-98.9 to 13.0] | -21.58 [-165.1 to 12.9]
  Week 12 | -9.40 [-114.9 to 17.6] | -15.00 [-188.3 to 50.5]
  Week 16 | -14.00 [-101.1 to 0.8] | -15.10 [-191.1 to 33.7]
  Week 20 | -9.50 [-108.5 to 0.1] | -12.80 [-194.2 to 21.5]
  Week 24 | -12.90 [-112.4 to 13.7] | -12.90 [-194.6 to 32.5]
  Week 26 | -11.20 [-103.4 to 16.8] | -6.90 [-194.6 to 22.5]

10. Secondary Outcome: Fecal Calprotectin: Change From Baseline (Week 0) to Week 8
Description: Stool samples for fecal calprotectin were collected before study drug administration when possible. Decreases in calprotectin are associated with decreased inflammation in the gastrointestinal tract. LOCF was used for missing data.
Time Frame: Baseline (Week 0) and Weeks 4 and 8
Population: ITT population.
Measure: Median (Full Range); unit: μg/g
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 15 | 15
μg/g
  Week 4 | -135.0 [-1441 to 3397] | -207.0 [-1334 to 3410]
  Week 8 | -44.0 [-1926 to 5632] | -274.0 [-915 to 6213]

11. Other Pre Specified Outcome: Number of Subjects Positive for Anti-Adalimumab Antibodies (AAA) From Baseline to Week 8
Description: Serum samples with adalimumab concentration below 2 μg/mL were selected for AAA analyses. Samples were considered AAA positive if the measured AAA concentration was above 2 μg/mL. A subject was considered to be AAA positive if the subject had at least one AAA positive sample observed within 30 days following the subject's last adalimumab dose. No samples were tested because all samples had adalimumab concentrations >2 μg/mL.
Time Frame: Baseline (Week 0) to Week 8
Population: ITT population.
Arm/Group | Low Induction Dose | Standard Induction Dose
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 35 weeks); SAEs were collected from the time informed consent was obtained (39 weeks).
Description: A TEAE in the double blind (DB) period is defined as any AE from the first dose of DB adalimumab to the first dose of open-label extension (OLE) adalimumab or 70 days after the last dose (for participants who did not enter OLE). A TEAE in the OLE period is any AE from the first dose of OLE adalimumab to 70 days after the last dose of study drug.
Groups:
- Low Induction Dose (Double-blind): Participants received the low loading dose of adalimumab (80 mg at Week 0) followed by the standard maintenance dose of adalimumab (40 mg every other week) at Weeks 2, 4, and 6.
- Standard Induction Dose (Double-blind): Participants received the standard loading dose of adalimumab (160 mg at Week 0 and 80 mg at Week 2) followed by the standard maintenance dose of adalimumab (40 mg every other week) at Weeks 4 and 6.
- Low Induction Dose (Open-label Extension); Standard Induction Dose (Open-label Extension): Participants received open-label adalimumab 40 mg every other week for 18 weeks.
Arm/Group | Low Induction Dose (Double-blind) | Standard Induction Dose (Double-blind) | Low Induction Dose (Open-label Extension) | Standard Induction Dose (Open-label Extension)
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 1/13 | 2/14
Other Adverse Events (participants affected / at risk) | 6/15 | 7/15 | 6/13 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Induction Dose (Double-blind) (N=15) | Standard Induction Dose (Double-blind) (N=15) | Low Induction Dose (Open-label Extension) (N=13) | Standard Induction Dose (Open-label Extension) (N=14)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 1 | 0 | 2
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
LUNG INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
TUBERCULOSIS GASTROINTESTINAL (Infections and infestations) | 0 | 1 | 0 | 0
MYCOBACTERIUM TUBERCULOSIS COMPLEX TEST POSITIVE (Investigations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Induction Dose (Double-blind) (N=15) | Standard Induction Dose (Double-blind) (N=15) | Low Induction Dose (Open-label Extension) (N=13) | Standard Induction Dose (Open-label Extension) (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 1 | 2 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ANAL ULCER (Gastrointestinal disorders) | 0 | 1 | 0 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ENTERITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
REGURGITATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ASTHENIA (General disorders) | 0 | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 0
PYREXIA (General disorders) | 2 | 1 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
GASTROINTESTINAL INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
VULVOVAGINAL INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
ACID BASE BALANCE ABNORMAL (Investigations) | 0 | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 0 | 1
CLOSTRIDIUM TEST POSITIVE (Investigations) | 0 | 1 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 1 | 0 | 0
MYCOBACTERIUM TUBERCULOSIS COMPLEX TEST POSITIVE (Investigations) | 0 | 0 | 0 | 2
PLATELET COUNT DECREASED (Investigations) | 0 | 1 | 0 | 0
RED BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1 | 0 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1 | 0 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
PHARYNGEAL ULCERATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.